CLINICAL TRIAL: NCT03093025
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study of the Safety and Efficacy of TS-121 as an Adjunctive Treatment for Patients With Major Depressive Disorder With an Inadequate Response to Current Antidepressant Treatment
Brief Title: A Study to Evaluate the Safety and Efficacy of TS-121 as an Adjunctive Treatment for Major Depressive Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Taisho Pharmaceutical R&D Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TS121-US201
Record Dates: First submitted 2017-03-15; First posted 2017-03-28 (Actual); Results first posted 2019-12-09 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Adjunctive Treatment
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TS-121 10mg (Experimental)
  Interventions: Drug: TS-121 10 mg
- TS-121 50mg (Experimental)
  Interventions: Drug: TS-121 50 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TS-121 10 mg — Orally taken once daily
  Arms: TS-121 10mg
Drug: TS-121 50 mg — Orally taken once daily
  Arms: TS-121 50mg
Drug: Placebo — Orally taken once daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of TS-121 as an adjunctive treatment for patients with major depressive disorder with an inadequate response to current antidepressant Treatment (SSRI, SNRI or bupropion).

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females between 18 and 65 years of age inclusive (at time of initial informed consent)
2. Patients with a current diagnosis of MDD by DSM-5, confirmed through a structured interview using MINI
3. Patients who receive the same antidepressant (SSRI, SNRI or bupropion monotherapy) for at least 6 weeks of continuous treatment with at least 4 weeks on a fixed dose
4. Patients who willing to remain on the same primary SSRI, SNRI or bupropion and fixed dose throughout the course of the study
5. Patients who meet the total score on the HAM-D as listed below

   1. HAM-D ≥ 18 at Screening
   2. HAM-D ≥ 18 at Baseline
6. Body Mass Index (BMI) ≥ 18 and ≤ 38 kg/m2

Exclusion Criteria:

1. Patients with inadequate response to ≥2 prior antidepressant treatments (not including current antidepressant) of at least 4 weeks duration each for the current episode
2. Patients whose current depressive episode is diagnosed with psychotic features, catatonic features, post-partum (primary onset), or is secondary to a general medical disorder
3. Patients with a diagnosis of any of the following DSM-5 class disorders

   1. Schizophrenia spectrum and other psychotic disorders
   2. Bipolar and related disorders
   3. Anxiety disorders [Co-morbid GAD and SAD will be allowed in the study if the primary diagnosis is MDD, and if in the opinion of the investigator, the comorbid anxiety is not likely to interfere with the subject's ability to participate in the trial or affect study outcome]
   4. Obsessive-compulsive and related disorders
   5. Trauma- and Stressor-related disorders
4. Patients who received electroconvulsive therapy (ECT) within 12 months of Screening, received more than one course of ECT in their lifetime or plan to receive ECT during the study
5. Patients who received repetitive transcranial magnetic stimulation (rTMS) within 12 months of Screening or plan to receive rTMS during the study
6. Patients who plan to initiate or terminate cognitive or behavioral psychotherapy or alter the frequency of ongoing therapy during this study
7. Patients who have attempted suicide within the past 6 months
8. Patients with history or presence of intellectual disability, pervasive developmental disorder, cognitive disorder, neurodegenerative disorder, or brain injury
9. Patients with any history or complication of convulsive disorder
10. Patients who are undergoing treatment with psychotropic medications, benzodiazepines, metyrapone, lithium and/or corticosteroids
11. Patients who are taking moderate to strong CYP3A4 inhibitors/inducers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2018-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shoji Yasuda, Study Chair — Taisho Pharmaceutical R&D Inc.
Locations (22):
- United States (22):
  - Woodland International Research Group, Little Rock, Arkansas
  - Woodland Research Northwest, Rogers, Arkansas
  - Collaborative Neuroscience Network, Garden Grove, California
  - PAREXEL Early Phase Clinical Unit, Glendale, California
  - Synergy East, Lemon Grove, California
  - NRC Research Institute, Orange, California
  - MCB Clinical Research Centers, Colorado Springs, Colorado
  - Comprehensive Psychiatric Care, Norwich, Connecticut
  - Compass Research, Orlando, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Chicago Research Center, Chicago, Illinois
  - Alexian Brothers Behavioral Health Hospital, Hoffman Estates, Illinois
  - Boston Clinical Trials, Boston, Massachusetts
  - Midwest Research Group - St. Charles Psychiatric Associates, Saint Charles, Missouri
  - St. Louis Clinical Trials, St Louis, Missouri
  - Hassman Research Institute, Berlin, New Jersey
  - Global Medical Institutes, Princeton, New Jersey
  - SPRI Clinical Trials, Brooklyn, New York
  - Midwest Clinical Research Center, Dayton, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Grayline Clinical Drug Trials, Wichita Falls, Texas

REFERENCES:
- [Background] Kamiya M, Sabia HD, Marella J, Fava M, Nemeroff CB, Umeuchi H, Iijima M, Chaki S, Nishino I. Efficacy and safety of TS-121, a novel vasopressin V1B receptor antagonist, as adjunctive treatment for patients with major depressive disorder: A randomized, double-blind, placebo-controlled study. J Psychiatr Res. 2020 Sep;128:43-51. doi: 10.1016/j.jpsychires.2020.05.017. Epub 2020 May 31. PMID 32521250
- See also: Related Info — https://doi.org/10.1016/j.jpsychires.2020.05.017

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TS-121 10mg | TS-121 50mg | Placebo
Started | 16 | 17 (One participant did not take any dose of investigational product after randomization.) | 18
Completed | 12 | 15 | 16
Not Completed | 4 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TS-121 10mg | TS-121 50mg | Placebo | Total
Number analyzed (Participants) | 16 | 16 | 18 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (12.62) | 44.8 (12.93) | 45.8 (11.09) | 45.1 (11.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 12 | 33
  Male | 6 | 5 | 6 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 4 | 3 | 13
  White | 7 | 10 | 12 | 29
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: The MADRS is a clinician-rated scale to assess depressive symptoms which consists from 10 items. The time frame for this scale is the past 7 days. Each item is scored on 7-point scale (0 [absence of symptoms] to 6 [severe]). The total score is the sum of 10 items and can take range from 0 to 60. A negative change from baseline indicates improvement.
Time Frame: 6 weeks
Population: Participants who did not receive at least one dose of investigational product or did not have at least one post-dose assessments were not included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TS-121 10mg | TS-121 50mg | Placebo
Number analyzed (Participants) | 13 | 15 | 17
score on a scale | -9.0 [-13.9 to -4.1] | -9.0 [-13.4 to -4.5] | -6.4 [-10.7 to -2.2]

2. Secondary Outcome: Hamilton Anxiety Scale (HAM-A)
Description: The HAM-A is a clinician-rated scale to assess anxiety symptoms which consists from 14 items. The time frame for this scale is the past 7 days. Each item is scored on 5-point scale (0 [absence of symptoms] to 4 [severe]). The total score is the sum of 14 items and can take range from 0 to 56. A negative change from baseline indicates improvement.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TS-121 10mg | TS-121 50mg | Placebo
Number analyzed (Participants) | 13 | 15 | 17
score on a scale | -5.6 [-8.1 to -3.1] | -3.4 [-5.7 to -1.2] | -2.8 [-5.0 to -0.6]

3. Secondary Outcome: Symptoms of Depression Questionnaire (SDQ)
Description: The SDQ is a self-rated scale to assess the severity of symptoms across several subtypes of depression which consists from 44 items. The time frame for this scale is the past 7 days. Each item is scored on 6-point scale (1 [better than normal] to 6 [severe]). The total score is the sum of 44 items and can take range from 44 to 264. A negative change from baseline indicates improvement.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TS-121 10mg | TS-121 50mg | Placebo
Number analyzed (Participants) | 13 | 15 | 17
score on a scale | -22.5 [-34.1 to -11.0] | -17.0 [-27.5 to -6.5] | -13.7 [-23.8 to -3.7]

4. Secondary Outcome: Clinical Global Impression-Severity (CGI-S)
Description: The CGI-S is a clinician-rated scale to assess the severity of the disorder. The time frame for this scale is the past 7 days. The score ranges from 1 (Normal, not ill at all) to 7 (Among the most extremely ill patients).
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TS-121 10mg | TS-121 50mg | Placebo
Number analyzed (Participants) | 13 | 15 | 17
score on a scale | -0.8 [-1.4 to -0.3] | -0.7 [-1.2 to -0.2] | -0.5 [-1.0 to 0.0]

5. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Percentage of MADRS responders (≥ 50% reduction in total score) at Week 6
Time Frame: 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | TS-121 10mg | TS-121 50mg | Placebo
Number analyzed (Participants) | 12 | 15 | 16
percentage of participants | 33.3 | 20.0 | 12.5

6. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I)
Description: Percentage of CGI-I improvers ("Very much improved" or "Much improved") at Week 6
Time Frame: 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | TS-121 10mg | TS-121 50mg | Placebo
Number analyzed (Participants) | 12 | 15 | 16
percentage of participants | 33.3 | 26.7 | 18.8

ADVERSE EVENTS:
Time Frame: Onset date on or later than date of first dose of the randomized treatment through follow-up visit, an average of 8 weeks.
Description: One participant in TS-121 50 mg group did not take any dose of investigational product after randomization. Therefore, the participant was not included in analyses.
Arm/Group | TS-121 10mg | TS-121 50mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/18
Other Adverse Events (participants affected / at risk) | 7/16 | 7/16 | 8/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TS-121 10mg (N=16) | TS-121 50mg (N=16) | Placebo (N=18)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Lenticular opacities (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoid infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bacterial test positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Crystal urine present (Investigations) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/25/NCT03093025/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/25/NCT03093025/SAP_001.pdf